CLINICAL TRIAL: NCT06083428
Title: Erector Spinae Plane Block (ESPB) vs. PENG Block for Pain Management and Stress Response in Patients Undergoing Total Hip Arthroplasty. A Prospective, Randomized Trial.
Brief Title: Erector Spinae vs. PENG Block for Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11/2023
Record Dates: First submitted 2023-05-24; First posted 2023-10-16 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hip Arthropathy; Hip Osteoarthritis; Hip Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG Block group (Active Comparator): ultrasound guided PENG block - 20ml 0,2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution - PENG block
- ESPB group (Active Comparator): ultrasound guided erector spinae plane block - 20ml 0,2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution Erector Spinae Plane Block
- Control group (Active Comparator): Only spinal anesthesia - No peripheral nerve block
  Interventions: Drug: Control Test

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution Erector Spinae Plane Block — ultrasound guided ESPB - L4 level, unilateral
  Other Names: Erector Spinae Plane Block
  Arms: ESPB group
Drug: Ropivacaine 0.2% Injectable Solution - PENG block — ultrasound guided PENG block
  Other Names: PENG block
  Arms: PENG Block group
Drug: Control Test — Only spinal anesthesia
  Other Names: No peripheral nerve block
  Arms: Control group

SUMMARY:
Effect of PENG block and ESPB on pain management, and NLR and PLR following knee arthroplasty

DETAILED DESCRIPTION:
Hip arthroplasty is one of the most common orthopedic procedures, especially in elderly patients, due to the deformation of joints. Patients may complain of severe pain due to surgical trauma and prosthesis. Regional anesthesia methods may be performed to reduce the inflammatory response, opioid consumption, and opioid-related side effects.

In recent years, the influence of regional anesthesiology on reducing the inflammatory response after surgical procedures has been emphasized. However, very few studies have evaluated the effect of various methods of anesthesia on the NLR.

This is the first study to investigate the effect of regional anesthesia on the NLR and PLR in patients undergoing hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III, Aged 20-90 years, Who will be scheduled for hip arthroplasty under spinal anesthesia.

Exclusion Criteria:

* Patients who have a history of bleeding diathesis, Take anticoagulant therapy, have a History of chronic pain before surgery, have Multiple trauma, cannot assess their pain (dementia), have been operated on under general anesthesia, have an infection in the area and do not accept the procedure

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 48 hours after surgery
  Total opiate consumption after surgery

SECONDARY OUTCOMES:
first need of opiate | 48 hours after procedure
  Time after surgery when the patient needs opiate for the first time
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 18 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 36 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Neutrophil-to-lymphocyte ratio | 24 hours after surgery
  Neutrophil-to-lymphocyte ratio
Neutrophil-to-lymphocyte ratio | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
Platelet-to-lymphocyte ratio | 24 hours after surgery
  Platelet-to-lymphocyte ratio
Platelet-to-lymphocyte ratio | 48 hours after surgery
  Platelet-to-lymphocyte ratio
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | Postoperative 24 hours period
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Domagalska, Ph.D., Principal Investigator — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No